CLINICAL TRIAL: NCT03513094
Title: The Effect of Volitional Transversus Abdominis Contraction on Time to Peak Sagittal Ground Reaction Force in Patients With Knee Osteoarthritis
Brief Title: Effect of TA Contraction on Gait in Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Daniel W. Flowers, Instructor of Physical Therapy, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 768
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Kinetics; Transversus abdominis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single group, repeated measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Without and With Transversus Abdominis (Experimental): Without:
  Participants performed three trials of self-selected, comfortable paced walking in the motion lab to collect kinetic data, without transversus abdominis contraction.
  With:
  Participants performed three trials of self-selected, comfortable paced walking in the motion lab to collect kinetic data, with 50% MVIC transversus abdominis contraction.
  Interventions: Other: Transversus Abdominis Contraction

INTERVENTIONS:
Other: Transversus Abdominis Contraction — Participants were educated on how to contract their transversus abdominis (TA) muscle after having a surface EMG biofeedback device placed on their abdomen to provide audible biofeedback. Participants were asked to ambulate while maintaining TA contraction while ambulating at 50% of maximal volitional isometric contraction.

SUMMARY:
The purpose of this study is to study the effects of core activation on knee joint loading during ambulation in patients with knee osteoarthritis (OA). This study aims to investigate the effects of transversus abdominis (TA) activation during simultaneous kinetic analysis of time to initial peak ground reaction force (T1) at the heel in the sagittal plane.

The objective of this study is to determine whether patients with knee OA demonstrate changes in T1 during comfortable gait speeds when actively contracting the TA muscle. In addition, this study will serve as a pilot study in order to perform a post-hoc power analysis for future study on the effects of the independent variable (TA contraction/changes in core stability) on the dependent variable (T1).

Null hypothesis: There will be no change in T1 in patients with knee OA during gait while contracting their TA.

Alternate hypothesis: There will be a decrease in T1 in patients with knee OA during gait while contracting their TA.

DETAILED DESCRIPTION:
This will be the first study on this topic performed by the investigator. Regarding current knowledge gaps, evidence has shown an influence of core strength measures/stability on lower extremity function. This relationship has been examined very little in patients with knee OA; however, evidence does show a correlation exists. There have been no studies examining the effect of a core strengthening/stability intervention on lower extremity kinetics in patients with knee OA to the PIs knowledge.

This is the first study examining the effects of TA contraction knee loading during gait in this population.

Current evidence shows that core activation/stability may play a role in lower extremity kinetics and kinematics. Most research has focused on younger, more athletic individuals. Research on this population has in the past looked at patellofemoral disorders or ligamentous injury. For example, decreased core function has been shown to increase the risk of sustaining anterior cruciate ligament injury. In addition, increased core stability has resulted in decreased knee loading during athletic activities.

There continues to be an overall paucity of research on proper prescription and dosage of therapeutic exercise for patients with knee OA. Evidence has shown that quadriceps strengthening and aerobic conditioning do lead to decreased disability. Additionally, patients with knee osteoarthritis have decreased postural stability as compared to healthy controls, with a significant correlation being observed between their score on a postural stability measure and the Western Ontario and McMaster Universities Osteoarthritis Index. Patients with knee OA also exhibit decreased overall core stability as compared to healthy controls. This body of research however does not include any evidence on the effects of a core stability intervention on improving overall function.

Knee OA leads to abnormalities in kinetic loading of the lower extremity during ambulation. An increase in T1 in this population has been observed when comparing to healthy controls. Separately, studies have shown that in patients with knee OA, knee joint loading can be influenced by intraarticular hyaluronic acid injections, resulting in decreased T1. Therefore, this study will explore the idea of how activation of a muscle (TA), which plays a large role in core stability, influences kinetic loading (T1) during ambulation in patients with knee OA.

Each participant will only be required to participate for one session, lasting about 1 hour. This does not included the informed consent process requiring approximately 30 minutes of their time prior to participation. Approximately 5 months will be required to enroll all participants. It is the PI's goal to complete primary data analysis no more than 3 months after data collection is complete, so total estimated study time is 8 months.

The primary study endpoint will be the cessation of data collection and the participants' active participation in the research program. The Secondary endpoint will be the completion of data analysis, which concludes the management of PHI.

Primary (exposure to any physical risk) and secondary (management of PHI) safety endpoints are synonymous with the study endpoints mentioned in 8.1.

This project serves as pilot study for future investigation on the role of core stabilization on gait kinetics in patients with knee OA. Therefore the sample size will be small. Post-hoc power analysis will inform the PI about requirements for participant recruitment needs for future investigations.

After informed consent is completed, participants will be scheduled for a session in the Motion Analysis Laboratory in the SAHP. Patients will have already been asked to wear close fitting, exercise appropriate clothing to allow marker placement, and prevent marker blocking during motion analysis. Data collection will begin by collecting the following anthropometric data: body weight (pounds, converted to kilograms) via a scale, height (inches, converted to mm) via a tape measure, leg length from ipsilateral anterior superior iliac spine to ipsilateral medial malleolus bilaterally (cm) via tape measure, and knee and ankle joint widths (cm) via a caliper. After collection of this data is completed and recorded, the PI will place reflective markers on the patient's skin via adhesive tape made for this purpose at the following landmarks bilaterally: ASIS, posterior superior iliac spine, lateral thigh, knee center of rotation, lateral leg, heel, lateral malleolus, and base of the second metatarsal. When this set-up is complete, static calibration of the motion analysis system will take place with the participant standing still in the capture area. When this is complete, the participant will be allowed a 2-minute warm-up by walking back and forth in the capture area. When this is completed the participant will be asked to walk at a comfortable pace across the capture area. Three trials with good force plate contact will be collected. After these three trials are obtained, the patient will lie supine on the mat in the lab, and will be taught how to perform a TA contraction. A Pathway MR-20 biofeedback device (The Prometheus Group, Dover, NH, USA) with two electrodes will be placed just medial to the ASISs on the participant's abdomen. A baseline maximal contraction will be performed supine, and the amplitude of contraction will be considered maximal voluntary isometric contraction (MVIC). The device will be set to provide audible feedback at 50% MVIC. The task will be repeated seated, standing, then ambulating three practice trials on the capture area. The participant will then be instructed to perform an additional three comfortable paced ambulation trials with good force plate contact while contracting the TA enough to cause audible feedback via the biofeedback device. After completing these three trials, the biofeedback device and reflective markers will be removed, and the participant will have completed their active participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* those with medical diagnosis (providing written evidence from a physician, physician assistant, or nurse practitioner) of knee OA unilaterally or bilaterally.

Exclusion Criteria:

* bilateral total knee arthroplasty, requirement of an assistive device or assistance with ambulation, spinal diagnoses which contraindicate participation in spinal stabilization activities, and those currently limited by another lower extremity pathology at the time of participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Kinetic Variable | During walking trials
  Time to first peak ground reaction force in the sagittal plane

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Flowers, DPT, Principal Investigator — LSUHSC-Shreveport
Locations (1):
- Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whyte EF, Richter C, O'Connor S, Moran KA. Effects of a dynamic core stability program on the biomechanics of cutting maneuvers: A randomized controlled trial. Scand J Med Sci Sports. 2018 Feb;28(2):452-462. doi: 10.1111/sms.12931. Epub 2017 Jul 13. PMID 28605148
- [Background] Messier SP, Loeser RF, Hoover JL, Semble EL, Wise CM. Osteoarthritis of the knee: effects on gait, strength, and flexibility. Arch Phys Med Rehabil. 1992 Jan;73(1):29-36. PMID 1729969
- [Background] Willson JD, Dougherty CP, Ireland ML, Davis IM. Core stability and its relationship to lower extremity function and injury. J Am Acad Orthop Surg. 2005 Sep;13(5):316-25. doi: 10.5435/00124635-200509000-00005. PMID 16148357
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] De Blaiser C, Roosen P, Willems T, Danneels L, Bossche LV, De Ridder R. Is core stability a risk factor for lower extremity injuries in an athletic population? A systematic review. Phys Ther Sport. 2018 Mar;30:48-56. doi: 10.1016/j.ptsp.2017.08.076. Epub 2017 Aug 24. PMID 29246794
- [Background] Shirey M, Hurlbutt M, Johansen N, King GW, Wilkinson SG, Hoover DL. The influence of core musculature engagement on hip and knee kinematics in women during a single leg squat. Int J Sports Phys Ther. 2012 Feb;7(1):1-12. PMID 22319676
- [Background] Ferber R, Bolgla L, Earl-Boehm JE, Emery C, Hamstra-Wright K. Strengthening of the hip and core versus knee muscles for the treatment of patellofemoral pain: a multicenter randomized controlled trial. J Athl Train. 2015 Apr;50(4):366-77. doi: 10.4085/1062-6050-49.3.70. Epub 2014 Nov 3. PMID 25365133
- [Background] Tang SF, Chen CP, Chen MJ, Pei YC, Lau YC, Leong CP. Changes in sagittal ground reaction forces after intra-articular hyaluronate injections for knee osteoarthritis. Arch Phys Med Rehabil. 2004 Jun;85(6):951-5. doi: 10.1016/j.apmr.2003.08.095. PMID 15179649
- [Background] Hsieh RL, Lee WC, Lo MT, Liao WC. Postural stability in patients with knee osteoarthritis: comparison with controls and evaluation of relationships between postural stability scores and International Classification of Functioning, Disability and Health components. Arch Phys Med Rehabil. 2013 Feb;94(2):340-6. doi: 10.1016/j.apmr.2012.09.022. Epub 2012 Oct 4. PMID 23041145
- [Background] Iversen MD. Managing Hip and Knee Osteoarthritis with Exercise: What is the Best Prescription? Ther Adv Musculoskelet Dis. 2010 Oct;2(5):279-90. doi: 10.1177/1759720X10378374. PMID 22870454
- [Background] Chen CP, Chen MJ, Pei YC, Lew HL, Wong PY, Tang SF. Sagittal plane loading response during gait in different age groups and in people with knee osteoarthritis. Am J Phys Med Rehabil. 2003 Apr;82(4):307-12. doi: 10.1097/01.PHM.0000056987.33630.56. PMID 12649658
- [Background] Roddy E, Zhang W, Doherty M. Aerobic walking or strengthening exercise for osteoarthritis of the knee? A systematic review. Ann Rheum Dis. 2005 Apr;64(4):544-8. doi: 10.1136/ard.2004.028746. PMID 15769914
- [Background] Daud DMBA, Razak NRA, Lasimbang H. CORE STABILITY DEFICITS IN FEMALE KNEE OSTEOARTHRITIS PATIENTS. Academic Journal of Science. 4(3):117-124, 2015.
- [Background] Dabholkar TA. Correlation of the core stability measures with the hip strength and functional activity level in knee osteoarthritis. International Journal of Therapies and Rehabilitation Research. 5(5):37-43, 2016.

DOCUMENTS (1):
  • Study Protocol (2017-05-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT03513094/Prot_000.pdf